CLINICAL TRIAL: NCT06247527
Title: Integrating a Transdiagnostic Psychological Intervention In The Care For Adolescents And Youth With HIV In Kenya
Brief Title: Psychoeducation, Relaxation, PrOblem Solving, Activation, Cognitive Coping Therapy for Adolescents and Youth in HIV Care
Acronym: PROACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: University of Washington (Other); Johns Hopkins University (Other); Kenyatta National Hospital (Other Government)
Responsible Party: Principal Investigator, Dalton Wamalwa, Associate Professor, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH133261 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Depression, Anxiety; Trauma; HIV-1-infection
MeSH Terms: conditions — Depression; Anxiety Disorders; Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Masking Description: Providers and participants will know the assigned arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROACT group (Experimental): Participants in intervention clinics with at least mild psychological distress (having depressive, anxiety or trauma symptoms) will receive a brief, modular, transdiagnostic psychological intervention (PROACT) delivered by non-specialist health providers at the HIV clinic.
  Interventions: Behavioral: Psychoeducation, Relaxation, PrOblem solving, Activation, Cognitive coping Therapy
- Control group (Active Comparator): Participants in control clinics with at least mild psychological distress (having depressive, anxiety or trauma symptoms) will be enrolled in the study, and will receive the standard of care interventions available in the HIV clinic.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Psychoeducation, Relaxation, PrOblem solving, Activation, Cognitive coping Therapy — This is a brief transdiagnostic psychological intervention based on the trauma-focused cognitive behavioral therapy (TF-CBT) designed for delivery by non-specialist providers to adolescents and youth with psychological distress
  Other Names: PROACT; Trauma-focused Cognitive Behavioral Therapy
  Arms: PROACT group
Behavioral: Standard of care — Any intervention, including counseling, provided as a routine intervention at the HIV clinic selected as a control clinic
  Arms: Control group

SUMMARY:
The proposed PROACT study will test the effectiveness of a mental health intervention (psychotherapy) for multiple common mental health conditions (depressive, anxiety and trauma symptoms) among adolescents and youth with HIV in Kenya. The study will also evaluate key factors for successful intervention implementation and conduct an economic evaluation to inform future intervention scale-up.

DETAILED DESCRIPTION:
Depression, anxiety, and trauma are common mental disorders that disproportionately affect adolescents and youth with HIV (AYHIV), and are associated with antiretroviral treatment (ART) non-adherence and poor treatment outcomes. The integration of mental health services in HIV care for AYHIV is recommended, but is lacking due to few trained mental health providers, and lack of a well validated integration models. Transdiagnostic interventions based on cognitive behavioral therapy (CBT) and delivered by lay health workers are effective in addressing these mental health conditions and could potentially improve HIV treatment outcomes. Barriers to integration of these interventions in the care of AYHIV in sub-Saharan Africa include paucity of effectiveness data among AYHIV and the lack of adaptation to tailor implementation for the HIV care context, including the length of treatment (number and frequency of sessions) and the format of delivery. This proposal builds on the successful pilot of 'Psychoeducation, Relaxation, PrOblem solving, Activation, Cognitive coping Therapy' (PROACT), a brief, modular and transdiagnostic intervention for adolescents and youth with mild to moderate symptoms of depression and anxiety in Kenya that resulted in clinically significant reduction in symptoms. The intervention can be delivered in stand-alone modules either in person or by phone, making it particularly appropriate for AYHIV when school is in session. In this project, we propose to further adapt PROACT for the HIV care setting through a stakeholder engagement process with policymakers, mental health and adolescent HIV practitioners, and AYHIV. Using a hybrid 1 cluster randomized trial in 30 HIV clinics in Kenya, we will assess the effectiveness of PROACT in reducing depressive, anxiety and trauma symptoms 6 months and 12 months after enrolment, comparing 300 AYHIV with mild to moderate symptoms in intervention to 300 in control clinics. To inform the integration of the intervention in routine care, we will measure implementation outcomes including reach, fidelity and maintenance, and explore multilevel determinants influencing reach, fidelity and maintenance in mental health screening and management, acceptability of training by providers and satisfaction with services by AYHIV. We will also conduct an economic evaluation through a time-driven activity-based costing of the intervention's implementation activities within the 30 clinics in participating in the study to estimate the implementation costs from a patient and health system perspective.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or youth ages 16-24 years attending HIV clinic at selected site with at least mild psychological distress who is willing to join the study and capable of providing consent to receive the intervention

Exclusion Criteria:

* If any study procedure would put them at an increased risk or if their compliance with study procedures is not possible

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 6 months and 12 months
  Symptoms measured using the 9-item Patient Health Questionnaire. Scores range from 0 to 27. Higher scores indicate more severe depressive symptoms
Anxiety | 6 months and 12 months
  Symptoms measured using the 7-item Generalized Anxiety Disorder scale. Scores range from 0 to 21. Higher scores indicate more severe anxiety
Trauma symptoms for AYHIV <18 years | 6 months and 12 months
  Symptoms measured using the Child and Adolescent Trauma Screen. Scores range from 0 to 60. Higher scores indicate more severe trauma distress symptoms
Trauma symptoms for AYHIV ≥18 years | 6 months and 12 months
  Symptoms measured using the Post Traumatic Stress Disorder checklist for 5th edition of the Diagnostic and Statistical Manual of Mental Disorders. Scores range from 0 to 80. Higher scores indicate more severe trauma distress symptoms

SECONDARY OUTCOMES:
Viral suppression | 6 months and 12 months
  HIV viral load measured from abstracted clinic records and defined as viral load of <200 copies/ml

OTHER OUTCOMES:
Reach | Early implementation (3 months) and late implementation (12 months)
  Proportion of AYHIV in intervention versus control clinics routinely screened using the PHQ-2/PHQ-9 tool out of total AYHIV who should be screened; and proportion of AYHIV in intervention clinics with psychological distress enrolled in the psychological intervention
Implementation fidelity | Early implementation (3 months) and late implementation (12 months)
  Proportion of intervention clinics implementing PROACT with high fidelity. Assessed using a standardized checklist and self-report

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nairobi, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data collected from participants after publication upon request. Data will be provided in accordance with the applicable laws and regulations in the United States and Kenya, and following requirements as per the NOT-MH-14-015 on Data Sharing Expectations for NIMH-funded Clinical Trials. We will package our data in a user-friendly format to facilitate use by other investigators, with a codebook documenting all variable names and values. Common data elements will be used to the extent possible. Additionally, we will create a syntax file of all scoring algorithms for computed scales and strategies for identifying and managing missing data.
Supporting Information: Study Protocol
Time Frame: The protocol will be available upon publication by June 2024 and the IPD will be available after publication of relevant papers
Access Criteria: Upon request to the study Principal Investigator